CLINICAL TRIAL: NCT01928368
Title: A Randomized, Double-Blind, Placebo-controlled, Ascending, Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 282 in Healthy Subjects and Subjects With Mild Atopic Asthma
Brief Title: A First-in-Human, Double Blind, Single Dose Study in Healthy Subjects and Subjects With Mild Atopic Asthma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20110235
Record Dates: First submitted 2013-08-21; First posted 2013-08-23 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Mild asthma; Atopic asthma; Healthy volunteers; First-in-human
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm (Active Comparator)
  Interventions: Drug: AMG 282
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: AMG 282 Matching Placebo

INTERVENTIONS:
Drug: AMG 282 — Single dose either subcutaneously or intravenously on day 1.
  Arms: Experimental Arm
Drug: AMG 282 Matching Placebo — Single dose of matching AMG 282 placebo either subcutaneously or intravenously on day 1.
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to determine if a single dose of AMG 282 is safe in healthy subjects and subjects with mild atopic asthma.

DETAILED DESCRIPTION:
A single SC or IV dose administration of AMG 282 to healthy subjects and subjects with mild atopic asthma will exhibit an acceptable safety and tolerability profile within the dose ranges studied.

ELIGIBILITY:
Inclusion Criteria (All subjects)

* Is a current non-smoker, has not used any nicotine or tobacco containing products (including but not limited to: snuff, chewing tobacco, cigars, cigarettes, pipes, or nicotine patches) within the last 6 months, and cumulative smoking history is ≤10 pack years.
* Females must be of documented non-reproductive potential (ie, postmenopausal [see definition below]; OR history of hysterectomy; OR history of bilateral salpingectomy; OR history of bilateral oophorectomy).
* Body mass index (BMI) between ≥ 18.0 and ≤ 32.0 kg/m2 at screening. (Subjects with mild atopic asthma only)
* Documented history of mild, stable atopic asthma within 2 years of screening.
* Has used only inhaled short-acting β2-agonists (less than twice weekly) to treat asthma.
* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) > 70% predicted at screening.

Exclusion Criteria

(All subjects)

* History or evidence of a clinically significant disorder, condition or disease that, in the opinion of the Principal Investigator or Amgen medical monitor would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Subject has a history of residential exposure to tuberculosis without a documented history of prophylactic treatment of tuberculosis or subject has a positive purified protein derivative (PPD) or QuantiFERON test at screening. Subjects with a documented negative PPD or QuantiFERON test within 4 weeks prior to screening who have no known tuberculosis exposure and have not traveled to an area with tuberculosis do not need to have a test performed at screening.
* Has donated or lost ≥ 500 mL of blood or plasma within 8 weeks of administration of the first dose of IP.

Other criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Up to day 141
Incidence of abnormal clinically significant vital signs | Up to day 141
Incidence of abnormal clinically significant chemistry, hematology and urinalysis test results | Up to day 141
Incidence of abnormal clinically significant ECG results | Up to day 141
Incidence of anti-AMG 282 antibodies | Up to 1 year

SECONDARY OUTCOMES:
Determination of various PK parameters including tmax, AUClast and Cmax | Up to day 141

OTHER OUTCOMES:
Measurement of various pharmacodynamic biomarkers in subjects with mild atopic asthma | Up to day 141

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - Research Site, Cypress, California
  - Research Site, Aventura, Florida
  - Research Site, Lenexa, Kansas
  - Research Site, Raleigh, North Carolina
  - Research Site, Seattle, Washington

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com